CLINICAL TRIAL: NCT05269979
Title: Hip Fracture Prevention by Screening and Intervention of Elderly Women in Primary Health Care. 2001 - 2022
Brief Title: Hip Fracture Prevention Follow-up of Elderly Women in Primary Health Care
Acronym: HIP22
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kronoberg County Council (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LU40600
Record Dates: First submitted 2022-02-05; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Fragility Fracture
Keywords: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (the Vislanda district) (Experimental): 435 women living in Vislanda responded to a detailed survey and participated in physical exercise and received lifestyle advice on diet, smoking, walking and outdoor activities. Recommendations to use calcium and Vitamin D and do exercise at home by written instructions. Home visit by rehab team when needed. Group training with a physiotherapist. Gymnastics group and walking group. Walking aides and instructions of anti-slip protection. Home environment risk reduction was offered.
  Interventions: Behavioral: Prevention of hip fractures
- Control (the Tingsryd/Emmaboda districts) (No Intervention): 415 women living in Tingsryd and 395 women living in Emmaboda responded to the same detailed survey as the 435 women living in Vislanda.

INTERVENTIONS:
Behavioral: Prevention of hip fractures — Physical exercise and lifestyle advice on diet, smoking, walking and outdoor activities. Recommendations to use calcium and Vitamin D and do exercise at home by written instructions. Home visit by rehab team when needed. Group training with a physiotherapist. Gymnastics group and walking group. Walking aides and instructions of anti-slip protection. Home environment risk reduction was offered.
  Arms: Intervention (the Vislanda district)

SUMMARY:
Researchers plan a 2022 follow-up of medical records data to investigate fracture incidence and survival for 1248 women, born 1902-1931, in a comparative fracture prevention study with 435 participants from an intervention area and 813 participants from two control areas.

In 2022 researchers want to assess patient records data in intervention and control areas and compare A) Survival B) Risk factors for osteoporotic fractures (wrist, upper arm, vertebral, pelvic, hip) C) physical activity, exercise and drugs that affect fracture risk.

DETAILED DESCRIPTION:
Researchers plan a 2022 follow-up of medical records data to investigate fracture incidence and survival for 1248 women, born 1902-1931, in a comparative fracture prevention study with participants from an intervention area (Vislanda, n=435) and control areas (Emmaboda n=395 and Tingsryd (n=418). Fragility fracture prevalence after 40 years of age was 33% in the 1248 participants with mean age 79 years at baseline 2001.

Participants with 2-4 risk factors (age ≥80, body weight <60kg, previous fragility fracture or impaired rise-up ability) provided prospective data with FRAMO (FRActure and Mortality) Index as an outcome measure and this index identified 80% of hip, fragility fractures or death within a 2-year follow-up period.

Hip fracture incidence 2004-2005 was not significantly lower in the intervention area but the trend of the odds ratio (0.33) was in line with significantly fewer falls and improved recovery in the intervention area.

In 2022 researchers want to assess patient records data in intervention and control areas and compare A) Survival B) Risk factors for osteoporotic fractures (wrist, upper arm, vertebral, pelvic, hip) C) physical activity, exercise and drugs that affect fracture risk. Data analysis will be blinded for participation in intervention or control groups and statistical methods include Cox regression and Kaplan-Meier's survival analyzes. Birth cohort differences in outcomes will be analysed by using Lexi's diagrams.

ELIGIBILITY:
Inclusion Criteria:

Invitation letter was sent out to all women in three predefined geographical areas of south Sweden born 1902-1931

Exclusion Criteria:

Participants who themselves or their significant others did not read or understand Swedish were excluded.

Ages: 70 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1248 (Actual)
Dates: Start 2001-11 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Survival | Maximum 21 years of follow up (Participants were on average 79 years old (70 to 100 years) at study start)
  Days
Fragility fractures | Maximum 21 years follow up
  Dates
Hip fractures | Maximum 21 years follow up
  Dates

SECONDARY OUTCOMES:
Time from fragility fractures until death | Maximum 21 years follow up
  Days